CLINICAL TRIAL: NCT02936622
Title: Paclitaxel-coated Peripheral Stents Used in the Treatment of Femoropopliteal Stenoses
Acronym: XPEDITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-002
Record Dates: First submitted 2016-10-12; First posted 2016-10-18 (Estimated); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Peripheral Arterial Disease (PAD)
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Stent 1 (Experimental): Zilver® PTX Stent
  Interventions: Device: Zilver® Paclitaxel-Eluting Peripheral Stent
- Stent 2 (Experimental): Zilver® Paclitaxel-Eluting Peripheral Stent with slower-dissolving polymer-free paclitaxel coating
  Interventions: Device: Zilver® Paclitaxel-Eluting Peripheral Stent with slower-dissolving polymer-free paclitaxel coating
- Stent 3 (Experimental): Zilver® Paclitaxel-Eluting Peripheral Stent with higher-dose polymer-free paclitaxel coating
  Interventions: Device: Zilver® Paclitaxel-Eluting Peripheral Stent with higher-dose polymer-free paclitaxel coating

INTERVENTIONS:
Device: Zilver® Paclitaxel-Eluting Peripheral Stent — Paclitaxel belongs to the Taxane drug class and coated on the stent at a much lower dose than when administered as a chemotherapy agent.
  Arms: Stent 1
Device: Zilver® Paclitaxel-Eluting Peripheral Stent with slower-dissolving polymer-free paclitaxel coating — Paclitaxel belongs to the Taxane drug class and coated on the stent at a much lower dose than when administered as a chemotherapy agent.
  Arms: Stent 2
Device: Zilver® Paclitaxel-Eluting Peripheral Stent with higher-dose polymer-free paclitaxel coating — Paclitaxel belongs to the Taxane drug class and coated on the stent at a much lower dose than when administered as a chemotherapy agent.
  Arms: Stent 3

SUMMARY:
This randomized multi-center study is intended to compare different coatings on stents for treatment of lesions of the above-the-knee femoropopliteal artery.

ELIGIBILITY:
Inclusion Criteria:

* One de novo or restenosed artherosclerotic lesion with ≥ 50% diameter stenosis
* Symptoms of peripheral arterial disease (Rutherford 2-4)

Exclusion Criteria:

* Pregnant, breastfeeding, or planning to become pregnant in the next 5 years
* Less than 18 years old
* Medical condition or disorder that would limit life expectancy to less than 12 months or that may cause noncompliance with the protocol or confound the data analysis
* Previous stent in the study vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
The percent diameter stenosis within the study lesion evaluated by conventional angiography. | 6 months
  Percent diameter stenosis will be calculated by comparing the minimal lumen diameter to the average of the proximal and distal reference vessel diameters.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, Prof. Dr. med., Principal Investigator — Universitäts Herzzentrum Freiburg - Bad Krozingen
Locations (11):
- Germany (10):
  - Klinikum Hochsauerland, Arnsberg
  - Universitäts Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Krankenhaud Bucholz, Buchholz
  - St. Josefskrankenhaus Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - SRH Klinikum Karlsbad- Langensteinbach GmbH, Karlsruhe
  - Universitatsklinikum Leipzig AoR, Leipzig
  - MEDINOS Kliniken des Landkreises Sonneberg GmbH, Sonneberg
  - Marienhospital Stuttgart, Stuttgart
  - Uniklinikum Würzburg, Würzburg
- Auckland City Hospital, New Zealand, Auckland, New Zealand